CLINICAL TRIAL: NCT05235594
Title: Feasibility of Monitoring Cancer Patients With a Smart T-shirt: Protocol for the OncoSmartShirt Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Helle Pappot, Professor, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OncoSmartShirt
Record Dates: First submitted 2022-01-28; First posted 2022-02-11 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: Patient reported outcomes; Smart t-shirt; Wearable; Patient-generated health data; Biometric sensor technology; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Smart shirt (Experimental): The research intervention is, for all twenty patients, to wear a smart t-shirt connected to a smart phone throughout the day (preferably 8 hours pr day) for 2 weeks.
  Interventions: Device: Wearable sensor

INTERVENTIONS:
Device: Wearable sensor — The patients will be asked to wear a smart shirt. The shirt is designed with multiple sensors and electrodes fully embedded which engender 6 different measurement flows continuously. The smart t-shirt system is washable, and patients can wash and dry this t-shirt anytime, thus the shirt can be worn repeatedly.
  Other Names: ChronolifeTM Smart t-shirt; OncoSmartShirt

SUMMARY:
The study will assess the feasibility of using the ChronolifeTM smart t-shirt for home monitoring of vital parameters in cancer patients during their treatment course. This study will bring new insights to how wearables and biometric data can be used as a part of symptom recognition in cancer patients during treatment course in the quest of increasing patients' quality of life.

DETAILED DESCRIPTION:
Collecting biometric sensor data by wearables is an example of real-time patient-generated health data that can provide vital and detailed objective information about patients. This may have the potential to improve quality of oncological treatment and increase patients' quality of life.

Studies have shown that there may be a dissimilar perception on symptoms and side effects between patients and health care professionals. Wearables may help identifying symptoms earlier.

A new design of a wearable is a smart t-shirt. A smart t-shirt has sensors embedded in the fabric which generate measurement flows. This new tool provide more precise information without recall and reporting bias which may have the potential to lead to a better and more accurate cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Danish cancer patients ≥18 years in antineoplastic treatment at Department of Oncology Rigshospitalet Denmark
* Both patients in curative and palliative care will be eligible
* 10 cancer patients under 39 years
* 10 cancer patients over 65 years
* Able to read and speak Danish

Exclusion Criteria:

* Serious cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who could wear the smart t-shirt preferably 8 hours pr. day during the three weeks study period | 2 weeks
  To assess the feasibility of using the ChronolifeTM smart t-shirt based on the completion rate which is defined as the number of included patients using the smart t-shirt at least 12 hours pr. day during the three weeks study period.

SECONDARY OUTCOMES:
Technical feasibility | 2 weeks
  To assess technical feasibility in a Danish healthcare system including data acquisition rate and data completeness.

OTHER OUTCOMES:
Changes in heart rate | 2 weeks
  Changes in heart rate (beat per minute) will be presented descriptively.
Changes in skin temperature | 2 weeks
  Changes in skin temperature (°C) will be presented descriptively.
Changes in physical activity | 2 weeks
  Changes in physical activity (steps) will be presented descriptively.
Changes in respirations frequency | 2 weeks
  Changes in respirations frequency (respiration per minute) will be presented descriptively.
Changes in thoracic impedance | 2 weeks
  Changes in thoracic impedance (kOhm) will be presented descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Holländer-Mieritz, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steen-Olsen EB, Pappot H, Green A, Langberg H, Hollander-Mieritz C. Feasibility of Monitoring Patients Who Have Cancer With a Smart T-shirt: Protocol for the OncoSmartShirt Study. JMIR Res Protoc. 2022 Oct 3;11(10):e37626. doi: 10.2196/37626. PMID 36190744